CLINICAL TRIAL: NCT01522664
Title: A Phase I, Open-Label Study of the Safety and Pharmacokinetics of Escalating Doses of DEDN6526A in Patients With Metastatic or Unresectable Melanoma
Brief Title: A Study of DEDN6526A in Patients With Metastatic or Unresectable Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO27935
Record Dates: First submitted 2012-01-20; First posted 2012-01-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

ARMS (1):
- Single group (Experimental)
  Interventions: Drug: DEDN6526A

INTERVENTIONS:
Drug: DEDN6526A — Multiple ascending doses

SUMMARY:
This multicenter, open-label study will assess the safety and pharmacokinetics of DEDN6526A in patients with metastatic or unresectable melanoma. Cohorts of patients will receive escalating doses of DEDN6526A by intravenous infusion on Day 1 of each 21-day cycle. In the absence of disease progression or unacceptable toxicity, patients may continue to receive DEDN6552A for up to 17 cycles (1 year).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Histologically confirmed metastatic melanoma (AJCC stage IV) or unresectable melanoma (AJCC Stage III)
* Prior failure of >/= 1 prior treatment regimens for metastatic or unresectable melanoma due to disease progression or unacceptable toxicity and for whom no standard therapy is available
* Measurable disease according to RECIST criteria
* Adequate bone marrow, liver and renal function
* Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to use one highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception through the course of the study treatment and for 6 months after the last dose of study treatment

Exclusion Criteria:

* Treatment with cytotoxic or antibody based therapy within 21 days prior to first dose of study treatment, or with any other anti-cancer therapy within 5 half-lives of the therapy prior to first dose of study treatment
* Known active infection (including HIV and atypical mycobacterial disease, but excluding fungal infection of the nail beds)
* Current Grad >/= 2 toxicity (except alopecia or anorexia) from prior therapy
* Grade >/= 2 peripheral neuropathy
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapies (or recombinant antibody-related fusion proteins)
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control)
* Evidence of significant uncontrolled concomitant disease or disorder
* Pregnant or lactating women
* Prior treatment with any other antibody-drug conjugate (ADC) compound containing monomethyl auristatin E (MMAE) for the treatment of melanoma
* Previous participation in a clinical trial within 30 days of the day of first study drug administration (Cycle 1, Day 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | assessed on an ongoing basis and up to 90 days following last dose of study treatment
Maximum tolerated dose/dose-limiting toxicities | approximately one year after study start
Determination of recommended Phase II dose | approximately 2 years

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve | Pre-dose, 30 min. and 4, 24, 48 hours post-dose and Days 7, 10, 15, 17 Cycles 1-4, pre-dose and 30 min. post-dose Cycle 5 and every other cycle thereafter
Anti-therapeutic antibody (ATA) levels | Pre-dose Day 1 Cycles 1-4, and within 30 days post last dose
Tumor response (tumor assessments according to RECIST criteria) | up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (6):
- United States (4):
  - Los Angeles, California
  - Sarasota, Florida
  - Detroit, Michigan
  - Nashville, Tennessee
- Australia (2):
  - Camperdown, New South Wales
  - East Melbourne, Victoria

REFERENCES:
- [Derived] Sandhu S, McNeil CM, LoRusso P, Patel MR, Kabbarah O, Li C, Sanabria S, Flanagan WM, Yeh RF, Brunstein F, Nazzal D, Hicks R, Lemahieu V, Meng R, Hamid O, Infante JR. Phase I study of the anti-endothelin B receptor antibody-drug conjugate DEDN6526A in patients with metastatic or unresectable cutaneous, mucosal, or uveal melanoma. Invest New Drugs. 2020 Jun;38(3):844-854. doi: 10.1007/s10637-019-00832-1. Epub 2019 Aug 5. PMID 31385109